CLINICAL TRIAL: NCT01824160
Title: Pulmonary Artery Repair With Covered Stents
Acronym: PARCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G120188
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Stenosis; Pulmonary Regurgitation; Tetralogy of Fallot
MeSH Terms: conditions — Pulmonary Valve Stenosis; Pulmonary Valve Insufficiency; Tetralogy of Fallot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Repair of RV-PA Conduit Disruption (Other): Covered stenting of RV-PA conduit injury
  Interventions: Device: Repair of RV-PA Conduit Disruption

INTERVENTIONS:
Device: Repair of RV-PA Conduit Disruption — Repair of RV-PA Conduit Disruption

SUMMARY:
The Covered Cheatham-Platinum Stent (CCPS) is being study for repair of tears that occur in the pulmonary artery during dilation (enlargement) of a conduit (passageway) connecting the right ventricle of the heart to the pulmonary arteries. Patients undergoing replacement of their pulmonary valve by transcatheter technique Melody Valve) are at risk of developing such tears in the process of preparing the conduit to accept the new valve. In order to implant such a valve, the connection between the right ventricle and the pulmonary arteries often needs to be enlarged. High pressure balloons may be needed and these balloons can sometimes cause tears in or even rupture of the connecting conduit. Such tears can allow blood to flow into the chest and rarely this can lead to a life-threatening emergency. Experience suggests that such tears can be closed by implanting into the conduit a metallic stent with an outer covering, rebuilding the wall and allowing continuation of the valve implant.

DETAILED DESCRIPTION:
Recent clinical reports from multiple pediatric cardiology programs around the world indicate that the conduit can be repaired using such a stent. In the United States there are no commercially available, FDA approved, covered stents of the size required. The Covered Cheatham Platinum Stent (CCPS) manufactured by the NuMED Corporation of Hopkinton, New York has been used in Europe since 2003 and more recently in Canada. The CCPS device is not yet approved by the Food & Drug Administration (FDA). However, it has been used at many hospitals in the U.S. to repair Right Ventricle to pulmonary artery conduits under Emergency and Compassionate Use circumstances. The NuMED Covered Cheatham-Platinum Stent (CCPS) is currently being studied for use in other areas of the body. The investigators are now studying its use in RV-PA conduits. The use of the Covered Cheatham Platinum Stent in this research study is investigational.

Only patients found to have a conduit tear during a Melody Valve implant procedure will be eligible for inclusion into the trial. Implant technique is left to the catheterization physician. Clinical data obtained during the catheterization, before and after the CCPS implant will be studied in order to understand factors leading up to the tear and to evaluate how successful the CCPS is in repairing such defects. Melody valve implant patients are routinely seen for clinical and echocardiographic reevaluation 6 months after implant. Patients who have received a CCPS during their Melody valve procedure will likewise be seen. Results from their clinical evaluation will be reviewed to make sure that the presence of a CCPS does not diminish the effectiveness of the Melody valve. Finally, the catheterization angiograms and 6 month follow up echocardiograms will be reviewed by an independent expert to confirm the clinical readings.

ELIGIBILITY:
Inclusion Criteria:

Precatheterization Inclusion Criteria:

1. Patient meets institutional criterion for placement of Melody® TPV
2. Patient size adequate to receive Melody TPV® implantation via venous access using the Ensemble® Transcatheter Delivery System
3. RV-PA conduit original size > 16 mm diameter
4. Patient age between 10 and 75 years

Catheterization Inclusion Criteria:

a. Angiographic evidence for RV-PA conduit disruption including: dissection, aneurysm, pseudo-aneurysm, tears or rupture

* Recognition and treatment of conduit disruption may occur before, during or after implantation of the Melody® TPV
* Conduit disruption related to prior intervention, identified angiographically before conduit dilation is performed during the Melody® implant procedure, can be eligible for CCPS implantation and study inclusion

Exclusion Criteria:

Precatheterization Exclusion Criteria:

1. Patient size too small for transvenous placement of the Melody® TPV
2. Bloodstream infection, including endocarditis
3. Pregnancy
4. Prisoners and adults lacking the capacity to give consent

Catheterization Exclusion Criteria:

1. Conduit size is not suitable (too small or too large) for a Melody® TPV
2. Risk of coronary compression has been identified
3. Lack of angiographic evidence for RV-PA conduit disruption - Prophylactic use of study CCPS is prohibited
4. Vessel injury occurring in either the right or left branch pulmonary arteries -If injury to branch pulmonary arteries occurs during the catheterization and covered stent usage is indicated, Emergency Use guidelines must be employed

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ringel, MD, Principal Investigator — Johns Hopkins University
Locations (38):
- United States (38):
  - Loma Linda University Health, Loma Linda, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - Rady Children's Hospital and Health Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Memorial Healthcare System, Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Miami Children's Hospital, Miami, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Advocate Children's Hospital - Oak Lawn, Oak Lawn, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Congenital Heart Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - Sunrise Children's, Children's Heart Center, Las Vegas, Nevada
  - Children's Hospital of New York - Presbyterian, New York, New York
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital/University of Uta, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Delaney JW, Goldstein BH, Bishnoi RN, Bisselou KSM, McEnaney K, Minahan M, Ringel RE; PARCS Investigators. Covered CP Stent for Treatment of Right Ventricular Conduit Injury During Melody Transcatheter Pulmonary Valve Replacement. Circ Cardiovasc Interv. 2018 Oct;11(10):e006598. doi: 10.1161/CIRCINTERVENTIONS.118.006598. PMID 30354627

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Repair of RV-PA Conduit Disruption
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants receiving a Covered CP stent for repair of pulmonary artery injury
Arm/Group | Repair of RV-PA Conduit Disruption
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Successful Repair of Conduit Disruption
Description: Successfully cover a tear or disruption in a RV-PA conduit wall and prevent the development of rupture or bleeding into the mediastinum during additional enlargement of the conduit. Provide persistent conduit wall integrity.
  A severity of illness scale categorizes the degree of clinical illness at baseline to be compared to the remaining level of illness after placement of the Covered CP Stent (CCPS). We assess the number of participants with minimal level of illness (level 0 to 1) after CCPS placement.
  0 = No injury or conduit wall disruption
  1. = Contained disruption
  2. = Partially contained disruption
  3. = Uncontained conduit disruption
Time Frame: Implant of Covered Stent and 6 month follow up
Measure: Number; unit: participants
Arm/Group | Repair of RV-PA Conduit Disruption
Number analyzed (Participants) | 50
participants | 48

ADVERSE EVENTS:
Arm/Group | Repair of RV-PA Conduit Disruption
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repair of RV-PA Conduit Disruption (N=50)
Stent malposition (Cardiac disorders) | 1 (1) — Stent became dislodged and migrated into the pulmonary arteries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No